CLINICAL TRIAL: NCT01372631
Title: A Novel Optical Spectral Imaging System for Imaging Breast Tumor Margins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00028284; 5R01EB011574 (NIH)
Record Dates: First submitted 2011-06-12; First posted 2011-06-14 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
Keywords: Reduction mammoplasty; mastectomy; partial mastectomy; lumpectomy; breast conserving surgery; breast cancer
MeSH Terms: conditions — Breast Neoplasms

ARMS (3):
- Pressure assessment (Experimental): 30 patients undergoing lumpectomy, mastectomy or reduction mammoplasty will be enrolled to assess the ideal pressure that should be applied when taking optical measurements.
  Interventions: Device: miniature spectral imaging system; Device: Bench-top optical spectrometer
- Random and Systematic Errors (Experimental): 40 patients undergoing lumpectomy or mastectomy will be enrolled to assess the random and systematic errors of the miniature spectral imaging system.
  Interventions: Device: miniature spectral imaging system; Device: Bench-top optical spectrometer
- Sensitivity and Specificity Assessment (Experimental): 150 patient undergoing lumpectomy, mastectomy or reduction mammoplasty will be enrolled in order to determine the sensitivity and specificity of the miniature spectral imaging system.
  Interventions: Device: miniature spectral imaging system; Device: Bench-top optical spectrometer; Device: High resolution microendoscope

INTERVENTIONS:
Device: miniature spectral imaging system — Use of miniature spectral imaging system
Device: Bench-top optical spectrometer — Use of bench-top optical spectrometer
Device: High resolution microendoscope — Use of high resolution microendoscope
  Arms: Sensitivity and Specificity Assessment

SUMMARY:
The goal of this research is to further develop novel optical assay systems for intra operative assessment of tumor margins in partial mastectomy or mastectomy specimens.

DETAILED DESCRIPTION:
The goal of this research is to further develop novel optical assay systems for intra operative assessment of tumor margins in partial mastectomy or mastectomy specimens. We are seeking to establish the accuracy of first and second-generation prototypes of technologies utilizing optical spectroscopy for intra operative margin assessment in partial mastectomy or mastectomy specimens. The aims associated with this research are as follows, (1) to evaluate the device-tissue interface on reduction mammoplasty specimens from a total of 20 patients, (2) to assess random and systematic errors of the new miniature system on mastectomy specimens from a total of 40 patients (3) to test the sensitivity, and specificity of the miniature spectral imaging system for margin assessment on excised partial mastectomy or mastectomy specimens from a total of 150 patients undergoing breast conserving surgery.

Last patient's surgery took place in 2017 and recruitment remained open. Later the team encountered staffing issues; therefore the study status was updated to suspended. We recently made the decision to no longer attempt to enroll the remaining 2 subjects and focus on the data analysis only.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a reduction mammoplasty OR
* Patients undergoing a lumpectomy mastectomy for the treatment of an invasive or non-invasive breast malignancy
* Age > 18
* Clinically detectable disease either by physical examination or radiographic studies
* Patients of all ethnic and gender groups will be included. Protocol accrual will be reviewed annually to include a determination of minority and gender representation. If accrual demonstrates under-representation of any group with comparison to disease incidence in that group, appropriate measures will be undertaken to increase participation of patients of that minority or gender group
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients considered in "vulnerable" populations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2011-04; Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Identification of the optical signatures in breast tissue | Day of procedure (less than 10 minutes)

SECONDARY OUTCOMES:
Sensitivity and Specificity of the device | Day of procedure (less than 10 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Nimmi Ramanujam, Ph.D., Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided